CLINICAL TRIAL: NCT03565146
Title: Evaluation of the Efficacy and Safety of PiQo4 System for the Treatment of Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Focus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Focus-PiQo4 Pigmentation-17-01
Record Dates: First submitted 2018-06-10; First posted 2018-06-21 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2018-06

CONDITIONS: Pigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pigmentation (Experimental): Treatment of Pigmented Lesions Using PiQo4 Laser System
  Interventions: Device: PiQo4 Laser System

INTERVENTIONS:
Device: PiQo4 Laser System — PiQo4 Laser System for treatment of pigmented lesions

SUMMARY:
A total of at least 25 healthy subjects at a single site, aged 21-70 years old with congenital or acquired challenging/resistant, age/sun-related flat and benign facial pigmentation with or without hand pigmentation who wish to improve their skin appearance.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Female or Male
2. Age= 21-70 (Adults)
3. Fitzpatrick skin phototype = I-V
4. Congenital or acquired benign pigmentation on face with optional pigmentation on hand.
5. Presence of at least 4 lesions of similar pigmentation intensity in the treatment area, in diameters larger than 2 mm
6. Able to read, understand and provide written Informed Consent
7. Able and willing to comply with the treatment/follow-up schedule and requirements
8. Women of child-bearing potential are required to use a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, Implanon or other FDA-approved devices, or abstinence) during the course of the study
9. Willing to have digital photographs taken of the treatment area
10. Willing to refrain from using any prescription or over the counter topical creams used for the treatment of pigmentation (e.g., hydroquinone, retinoids, and/or corticosteroids) in the treatment area during the study period.
11. Willing to protect from sun exposure and use an approved sunscreen of SPF 30 or higher in the treatment area daily during the entire duration of the study, including the follow-up period.
12. Agree not to undergo any other procedure(s) for the treatment of pigmentation or solar lentigines during the study.

Exclusion Criteria:

1. History of post inflammatory pigmentary disorders, particularly a tendency for hyper- or hypo-pigmentation
2. Melasma
3. Excessive underlying vascular conditions (e.g. dense network of capillaries)
4. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 3 months after completion of breastfeeding
5. Prior skin laser, light, or other energy device treatment in treated area within 6 months of initial treatment or during the course of the study
6. Prior ablative resurfacing procedure or face-lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study
7. Prior treatment with medium-depth or deeper chemical peels or dermabrasion in treated area within 3 months of initial treatment or during the course of the study
8. Prior use of any prescription or over the counter topical creams used for the treatment of pigmentation (e.g., hydroquinone, retinoids, and/or corticosteroids) in the treatment area within 3 months of initial treatment or during the course of the study
9. Any other surgery in treated area within 9 months of initial treatment or during the course of the study
10. Hypersensitive to light exposure or the use of photosensitive medication for which light exposure is contraindicated
11. Multiple dysplastic nevi in area to be treated
12. Significant concurrent illness (e.g. uncontrolled diabetes) or any disease state that in the opinion of the Investigator would interfere with the treatment or healing process
13. Any dermal/epidermal damage or disorder, mainly vascular or textural lesions, in the treatment area.
14. Any underlying tattoo in the treatment area.
15. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study
16. Participation in a study of another investigational device or drug involving the same anatomical site within 3 months prior to enrollment or during this evaluation, or if not involving the same anatomical site, as per the Investigator's discretion
17. History of keloid or any other type of hypertrophic scar formation or poor wound healing
18. Signs and symptoms of hormonal disorders such as Melasma, as per the Investigator's discretion.
19. Concurrent inflammatory skin conditions, open laceration, or abrasion of any sort on area to be treated during the course of treatment
20. Active Herpes Simplex (perioral or facial) at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment
21. Having a bleeding disorder or taking anticoagulation medications, including daily use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to treatment (as per the discretion of the subject's primary care physician)
22. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or the use of immunosuppressive medications
23. Having any form of active cancer at the time of enrollment and during the course of the study or history of skin cancer on the face/hands
24. Pigmented lesions in the areas to be treated that are suspicious for pre-malignancy or malignancy and/or are not deemed suitable for phototherapy, as per the Investigator's discretion
25. Unable to understand or provide written Informed Consent (e.g. mental incompetence or evidence of active substance abuse)
26. Any condition that, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study
27. If undergoing punch biopsy, allergic to lidocaine or epinephrine

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Pigmentation Improvement Scale | 1 month follow up
  Facial Pigmentation Improvement evaluated by the investigator at the 1 month follow up visit compared to baseline using a 5-point improvement scale where a score of between 0 and 4 will be assigned (0-No improvement; 1- Trace to mild improvement of some lesions; 2- Moderate response: some lesions lighter; 3- Good response: most lesions much lighter; 4 - excellent response: most or all lesions are much lighter or gone)

SECONDARY OUTCOMES:
Pigmentation Improvement Scale | 3 month follow up
  Facial Pigmentation Improvement evaluated by the investigator at the 3 month follow up visit compared to baseline using a 5-point improvement scale where a score of between 0 and 4 will be assigned (0-No improvement; 1- Trace to mild improvement of some lesions; 2- Moderate response: some lesions lighter; 3- Good response: most lesions much lighter; 4 - excellent response: most or all lesions are much lighter or gone)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Friedmann, Principal Investigator — Westlake Dermatology
Locations (1):
- Westlake Dermatology, Austin, Texas, United States